CLINICAL TRIAL: NCT00533403
Title: MK0686 in Postsurgery Dental Pain (0686-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0686-002; 2007_617
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — methyl 3-chloro-3'-fluoro-4'-(1-(((1-((trifluoroacetyl)amino)cyclopropyl)carbonyl)amino)ethyl)-1,1'-biphenyl-2-carboxylate

INTERVENTIONS:
Drug: MK0686

SUMMARY:
To compare the pain relieving effect of MK0686 to placebo or ibuprofen after dental surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-45 years who are scheduled to have 2 or more third molars (wisdom teeth) removed
* Patients must agree to remain in the clinic for 24 hours after surgery

Exclusion Criteria:

* Patient has history of heart disease, asthma, pulmonary disease
* Patient must discontinue use of certain pain medicines 24-72 hours prior to the surgery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2004-07; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC